CLINICAL TRIAL: NCT05693454
Title: Local Wound Anesthesia in Spine Surgery - a Randomized Double Blind Controlled Trial
Brief Title: Local Wound Anesthesia in Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LAWS
Record Dates: First submitted 2021-07-20; First posted 2023-01-23 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Surgical Wound; Orthopedic Disorder of Spine
MeSH Terms: conditions — Surgical Wound | interventions — Tramadol

STUDY DESIGN:
Intervention Model Description: randomized, double blind, controlled
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): local wound infiltration at the end of spine surgery with NaCl
  Interventions: Drug: Infiltration with NaCl
- Arm I (Active Comparator): local wound infiltration at the end of spine surgery with Ropivacain
  Interventions: Drug: Infiltration with Ropivacain
- Arm II (Active Comparator): local wound infiltration at the end of spine surgery with a combination of Levobupivacaine and Tramadol
  Interventions: Drug: Infiltration with a combination of Levobupivacaine and Tramadol

INTERVENTIONS:
Drug: Infiltration with NaCl — Local wound infiltration at the end of spine surgery with NaCl
  Arms: Control
Drug: Infiltration with Ropivacain — Local wound infiltration at the end of spine surgery with Ropivacain
  Arms: Arm I
Drug: Infiltration with a combination of Levobupivacaine and Tramadol — Local wound infiltration at the end of spine surgery with a combination of Levobupivacaine and Tramadol
  Arms: Arm II

SUMMARY:
Prospective, randomized, double-blinded, trial regarding the effect of local wound infiltration at the end of spine surgery; randomizing 1:1:1 between NaCl, Ropivacain, Levobupivacaine combined with Tramadol

DETAILED DESCRIPTION:
Subcutaneous local wound injections with NaCl, Ropivacain or Levobupivacaine combined with Tramadol will be performed in a randomized, double-blinded manner at the end of spine surgery. Pain control, dosage of analgesics used, analgesics reduction compared to preoperative, wound healing problems and clinical outcome socres will be assessed up to 6 weeks after surgery

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Age ≥ 18 years
* Elective spine surgery with any technique
* At least 6 weeks of scheduled follow-up from hospitalization

Exclusion Criteria:

* Documented decline for data inclusion
* Allergy to any of the drugs used
* <50kg total body weight
* Vertebro- or Kyphoplasty
* Pregnancy and breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Pain control | 2 hours after surgery
  pain assessment by visual analog with 0 = no pain and 10 = maximal pain
Pain control | 4 hours after surgery
  pain assessment by visual analog with 0 = no pain and 10 = maximal pain
Pain control | 8 hours after surgery
  pain assessment by visual analog with 0 = no pain and 10 = maximal pain
Pain control | 12 hours after surgery
  pain assessment by visual analog with 0 = no pain and 10 = maximal pain
Pain control | until 42 days after surgery
  analgesics consumption

SECONDARY OUTCOMES:
costs | at 42 days after surgery
  total costs for the intervention under study in Swiss Francs
sick leave | at 42 days after surgery
  duration of sick leave
hospital stay | up to 8 weeks
  length of hospital stay in days
wound drying | up to 8 weeks
  time in days until wound is dry
wound length | up to 8 weeks
  wound length
wound healing | until 42 days after surgery
  have wound healing problems occurred (yes / no)

CONTACTS AND LOCATIONS:
Overall Officials: Mazda Farshad, Prof, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers outside of our institution